CLINICAL TRIAL: NCT01517022
Title: Impact of a Package of Intensive Smoking-cessation Interventions Versus Smoking-cessation Advice on Outcomes in Smear-positive Patients With Pulmonary Tuberculosis; a Randomised Controlled Trial (STB_RCT).
Brief Title: Intensive Smoking-cessation Intervention Versus Smoking-cessation Advice in Smear-positive Patients With Pulmonary Tuberculosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: University of Cape Town (Other); Sri Venkateswara Institute of Medical Sciences University (Other)
Responsible Party: Principal Investigator, S.K.SHARMA, Professor and Head, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SKS/Med/NI1161
Record Dates: First submitted 2011-06-23; First posted 2012-01-25 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Tuberculosis
Keywords: smoking cessation; early sputum smear conversion
MeSH Terms: conditions — Tuberculosis; Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control arm (No Intervention): Control arm patients will receive pre designed pamphlets and structured conselling for smoking cessation by trained counsellors along with routine DOTS treatment
- Intervention arm (Active Comparator): Cessation arm patients will receive pre designed pamphlets and structured conselling for smoking cessation by trained counsellors along and nicotine replacement therapy(NRT) and routine DOTS treatment
  Interventions: Drug: nicotine replacement therapy

INTERVENTIONS:
Drug: nicotine replacement therapy — nicotine replacement therapy 2mg for patients cessation arm for period of 6 weeks
  Other Names: Nicogum 2mg Cipla pharmaceuticals
  Arms: Intervention arm

SUMMARY:
The aim of the study is to determine the impact of a package of smoking-cessation interventions on a composite measure of Tuberculosis (TB) treatment-related outcomes.

Given the lack of objective clinical data/evidence about the impact of smoking-cessation on TB-related outcomes, yet subjective expert opinion that smoking cessation is highly likely to be beneficial particularly in patients with TB, this study proposes to determine the impact of an intensive package of smoking-cessation interventions aimed to promote smoking-cessation (counseling plus nicotine replacement therapy, NRT), on patient response to anti-tuberculosis therapy. This is to be compared with the structured counselling for smoking-cessation that is recommended to be routinely provided by health care workers to all patients who are smokers. If the results prove that such a smoking-cessation PI indeed improves outcomes in TB patients, such information would strongly motivate for the institution of more intensive smoking-cessation interventions in TB clinics than is currently being employed for TB patients

DETAILED DESCRIPTION:
No clinical trials have been done to determine if the cessation of smoking has any influence on outcome in tuberculosis patients. In particular, if smoking cessation leads to a higher rate of sputum culture-conversion at 2 months, TB transmission rates should be reduced. Such targeted smoking-cessation intervention may be more successful than general public education strategies in reducing the spread of TB in high-incidence countries Tuberculosis (TB) . The WHO has estimated that approximately a third of the world's population is infected with Mycobacterium tuberculosis, and approximately 2 million die from TB every year. Tobacco smoking, which is the single most preventable cause of death in the world today, appears to be an important risk factor for TB disease and mortality, especially in countries such as India. The smoking-TB association has major public health implications because in many of the developing countries where there is a high prevalence of TB, smoking is also a common practice. Smoking is widespread, with approximately a third of the global population aged 15 years or above being smokers, but has reached epidemic proportions in countries such as India, China and Russia. For example, in India more than half of the rural male population is estimated to smoke and India accounts for 1.85 million TB cases each year. Therefore in India, as for other developing countries, the co-existence of a high TB and smoking burden is a major health concern, and further underscores the importance of promoting smoking cessation to the general public. In India, studies have shown a strong association between tobacco and TB mortality. An estimated third of male TB deaths in India may be due to smoking. However, there is concern that many of the published studies did not adequately control for bias and confounding (that may have caused spurious associations).

ELIGIBILITY:
Inclusion Criteria:

* any adult (> 18 years)
* Recently diagnosed (primary TB/Relapse TB) smear-positive TB patient who self-reports to smoke at least 10 whole cigarettes or bidis (rolled tobacco leaf) per day, every day

Exclusion Criteria:

* patients will be excluded from recruitment to the study if they fall into any one or more of these exclusion categories:

  * Inability to give consent or < 18 years
  * Patients who self-report to smoke less than 10 whole cigarettes/bidis per day
  * TB patients who have already started anti-tuberculosis therapy for more than 1 week.
  * Patients with known multidrug-resistant TB (or XDR) (information provided by patient or the information is available in the clinic folder).
  * Known HIV-positive patients
  * Contra-indications to NRT (patients with a history of severe cardiovascular disease including arrhythmias, recent myocardial infarction (within the last 6 months), recent cerebrovascular incident (6 months), and/ or history of peripheral vascular disease, phaeochromocytoma, poorly controlled diabetes mellitus, hyperthyroidism, renal/hepatic impairment or gastritis/peptic ulcers). Patients with asthma or depression will also be excluded, as quitting may have an effect on medications used for these conditions. Patients with severe skin disorders (such as psoriasis or eczema) will also be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2010-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
1. Change in TB Score at second month and sixth month | Measured at baseline, second month and sixth month.
  Composite score for objective and subjective improvement measured at baseline, second month and sixth month
Sputum culture conversion | Measured at baseline and second month
  Sputum culture conversion at second month using solid/liquid culture technique

SECONDARY OUTCOMES:
Sputum smear conversion | Measured at baseline, second week, fourth week, second month and sixth months
  Protocol was amended to access sputum conversion weekly up to second month
Mortality at sixth month | Sixth month
  To determine number of mortality at the end of follow-up
More than 10% weight gain at six months | Sixth month
  To determine rate of weight gain after completion of treatment
Proportion of subjects in each group that have quit smoking at second month | Sixth month
  To determine the rate of smoking cessation in the cohort
Treatment completion | Six months for new cases and eight months for re-treatment cases following regimen 2
Cure, failure and default rate | At sixth month
  To determine cure, failure and default rate in the cohort

CONTACTS AND LOCATIONS:
Overall Officials: Surendra K Sharma, MD, Ph.D., Principal Investigator — AIIMS, New Delhi
Locations (1):
- All India Institute of Medical Sciences, Ansari Nagar, New Delhi, India

REFERENCES:
- [Derived] Hartmann-Boyce J, Theodoulou A, Farley A, Hajek P, Lycett D, Jones LL, Kudlek L, Heath L, Hajizadeh A, Schenkels M, Aveyard P. Interventions for preventing weight gain after smoking cessation. Cochrane Database Syst Rev. 2021 Oct 6;10(10):CD006219. doi: 10.1002/14651858.CD006219.pub4. PMID 34611902